CLINICAL TRIAL: NCT05568316
Title: Impact of Immunonutrition on Nutritional Status in Patients Undergoing Colorectal Cancer Surgery: A Randomised Controlled Clinical Trial
Brief Title: Impact of Immunonutrition on Nutritional Status in Colorectal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/151-2879
Record Dates: First submitted 2022-08-25; First posted 2022-10-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Immunonutrition; Nutritional Status
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Preoperative Immunonutrition (Group 1) (Experimental): Participants received oral IMN supplementation containing arginine, omega-3 fatty acids, and dietary nucleotides for only 5 days before surgery, in addition to their standard isocaloric diet.
  Duration: 5 days (preoperative) Dietary therapy: Standard oral nutrition and IMN product for 5 days before operation.
  The nutritional status of the patients was determined from the NRS 2002 screening tool. The biochemical parameters (albumin, prealbumin, CRP, FPG etc.), anthropometric measurements (body weight, BMI, MUAC), postoperative complications and hospital stay were recorded.
  Interventions: Dietary Supplement: Preoperative Immunonutrition
- Experimental: Perioperative Immunonutrition (Group 2) (Experimental): Participants received oral IMN supplementation containing arginine, omega-3 fatty acids, and dietary nucleotides for 5 days before and after surgery, in addition to their standard isocaloric diet.
  Duration: 5 days preoperative and 5 days postoperative Dietary therapy: Standard oral nutrition and IMN product for 5 days before and after operation (perioperative).
  The nutritional status of the patients was determined from the NRS 2002 screening tool. The biochemical parameters (albumin, prealbumin, CRP, FPG etc.), anthropometric measurements (body weight, BMI, MUAC), postoperative complications and hospital stay were recorded.
  Interventions: Dietary Supplement: Perioperative Immunonutrition

INTERVENTIONS:
Dietary Supplement: Preoperative Immunonutrition — Participants consumed oral IMN supplementation containing arginine, omega-3 fatty acids, and dietary nucleotides for 5 days before surgery.
  The nutritional status of patients was evaluated according to the score determined from the NRS 2002 screening tool. Anthropometric measurements (height, body weight, BMI, and middle-upper arm circumference) were measured at the beginning (7 days before the operation) and seventh day after the operation. The biochemical parameters (albumin, prealbumin, C-reactive protein, fasting plasma glucose, alanine aminotransferase, and aspartate aminotransferase) of participants were recorded 7 days before, on the day, and 7 days after the operation from hospital patients forms.Infections (such as urinary tract, wound infections), complications, and the length of patients' hospital stay were recorded during the postoperative period.
  Arms: Experimental: Preoperative Immunonutrition (Group 1)
Dietary Supplement: Perioperative Immunonutrition — Participants received oral IMN supplementation containing arginine, omega-3 fatty acids, and dietary nucleotides for 5 days before and after surgery, in addition to their standard isocaloric diet.
  The nutritional status of patients was evaluated according to the score determined from the NRS 2002 screening tool. Anthropometric measurements (height, body weight, BMI, and middle-upper arm circumference) were measured at the beginning (7 days before the operation) and seventh day after the operation. The biochemical parameters (albumin, prealbumin, C-reactive protein, fasting plasma glucose, alanine aminotransferase, and aspartate aminotransferase) of participants were recorded 7 days before, on the day, and 7 days after the operation from hospital patients forms.Infections (such as urinary tract, wound infections), complications, and the length of patients' hospital stay were recorded during the postoperative period.
  Arms: Experimental: Perioperative Immunonutrition (Group 2)

SUMMARY:
Colorectal cancer is among the top three types of cancer that are most common and causes death worldwide.Nutritional support is widely used in elective colorectal surgery patients, as nutritional status is an important factor affecting clinical outcomes. European Society for Clinical Nutrition and Metabolism (ESPEN, 2016) emphasizes that nutritional supplementation with compounds such as amino acids, arginine, glutamine, and fish oil (omega 3) improves postoperative recovery.

Glutamine; it becomes an essential amino acid under stress. It is an energy substrate for cells such as intestinal mucosal cells and lymphocytes, a material for glutathione synthesis, and a potent antioxidant, which also increases heat shock protein expression. In stressful conditions, arginine is the primary fuel source for T cells and is required for nitric oxide synthesis; therefore, it helps maintain immune function. Omega 3; It plays a role in the treatment of inflammation and improves wound healing. In addition, EPA and DHA increase the immune response by improving lymphocyte function. RNA; They are essential for maturation, proliferation, and function in nearly all biochemical processes, in rapidly proliferating cells such as T cells. studies have shown that immunonutrition (IMN) formulas enriched with biologically active compounds may be more effective in reducing infection complications and shortening postoperative hospital stays.

This study aimed to investigate the additional effects of perioperative compared with preoperative immunonutrition on anthropometric, nutritional, and biochemical parameters, complications, and the length of hospital stay in patients with colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is one of the five most common cancer types in men and women worldwide. Cancer malnutrition is seen in patients with colorectal cancer, and this adversely affects the prognosis of the disease. Major operations performed may lead to dysfunction in body homeostasis, impaired defense mechanisms and inflammatory response, increasing the risk of postoperative complications and prolonging hospital stay. Nutritional support products enriched with special compounds such as arginine, glutamine, and omega3 may contribute to the daily energy intake of patients, as well as support the immune system, increase wound healing, and reduce the risk of infection. It is well-documented that preoperative and perioperative compared to no immunonutrition effectively reduce the risk of developing infectious complications and the length of hospital stay. Unless, studies on this subject are very few, especially in our country, Turkey, and their results are contradictory.

The aim of this study is to investigate the additional effects of perioperative compared with preoperative immunonutrition (IMN) on anthropometric, nutritional, biochemical parameters, hospital stay and postoperative complication in patients with colorectal cancer.

The hypotheses of this study are as follows:

H0: There is no difference between the consumption of perioperative compared with preoperative immunonutrition (IMN) on anthropometric, nutritional, biochemical parameters, hospital stay and postoperative complication in patients with colorectal cancer.

H1: Perioperative immunonutrition compare to preoperative has a positive effect in improving the anthropometric measurements, nutritional and biochemical parameters, hospital stay and postoperative complication in patients with colorectal cancer.

Primary purpose: To evaluate the effects of IMN on anthropometric measurements, nutritional and biochemical values of participants in groups.

Secondary purpose: To evaluate the effects of IMN on postoperative complications and length of hospital stay in groups.

The study was conducted as a single-blind prospective randomized controlled clinical trial at a single institution, Haydarpasa Numune Training and Research Hospital General Surgery Clinic, Istanbul, Turkey, between November 2020 and October 2021. The participants included consecutive patients undergoing colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with colorectal cancer,
* from 18 years up to 65 years old,
* To be volunteer,
* Informed written consent

Exclusion Criteria:

* Under the age of 18,
* Above the age of 65
* To be pregnant,
* Acute and chronic renal failure, cirrhosis, advanced COPD, mechanical intestinal obstruction, metastasis, presence of sepsis,
* The ejection fraction is below 35%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Nutritional Status | At the beginning of the study (7 days before the operation)
  The nutritional status of patients was evaluated according to the score determined from the NRS 2002 screening tool. Score >3: The patient is at risk for nutrition and a nutrition facility is started Score <3: one should be scanned. If there is a major operation plan, a nutrition plan should also be developed.
Anthropometric Measurements | At the beginning of the study (7 days before the operation)
  Height in meters was measured by researchers at the begining of the study.
Anthropometric Measurements | At the beginning of the study (7 days before the operation)
  Body weight in kilogram was measured by researchers.
Anthropometric Measurements | At the beginning of the study (7 days before the operation)
  Weight and height will be combined to report BMI in kg/m^2
Anthropometric Measurements | At the beginning of the study (7 days before the operation)
  Middle-upper arm circumference (MUAC) in centimeter was measured by using tape measure.
Biochemical Measurements | At the beginning of the study (7 days before the operation)
  Albumin levels in g/dL of participants was recorded from hospital's patients form.
Biochemical Measurements | At the beginning of the study (7 days before the operation)
  Prealbumin levels in mg/dL of participants was recorded from hospital's patients form.
Biochemical Measurements | At the beginning of the study (7 days before the operation)
  Fasting plasma glucose (FPG) mg/dL in of participants was recorded from hospital's patients form.
Biochemical Measurements | At the beginning of the study (7 days before the operation)
  Alanine aminotransferase (ALT) in IU/L of participants was recorded from hospital's patients form.
Biochemical Measurements | At the beginning of the study (7 days before the operation)
  Aspartate aminotransferase (AST) in IU/L of participants was recorded from hospital's patients form.
Biochemical Measurements | At the beginning of the study (7 days before the operation)
  C-reactive protein (CRP) in mg/L of participants was recorded from hospital's patients form.
Anthropometric Measurements | 7th day after the operation
  Body weight in kilogram was measured by researchers.
Anthropometric Measurements | 7th day after the operation
  Weight and height will be combined to report BMI in kg/m^2
Anthropometric Measurements | 7th day after the operation
  Middle-upper arm circumference (MUAC) in centimeter was measured by using tape measure.
Biochemical Measurements | On the operation day (Day 0)
  Albumin levels in g/dL of participants was recorded from hospital's patients form.
Biochemical Measurements | On the operation day (Day 0)
  Prealbumin levels in mg/dL of participants was recorded from hospital's patients form.
Biochemical Measurements | On the operation day (Day 0)
  Fasting plasma glucose (FPG) mg/dL in of participants was recorded from hospital's patients form.
Biochemical Measurements | On the operation day (Day 0)
  Alanine aminotransferase (ALT) in IU/L of participants was recorded from hospital's patients form.
Biochemical Measurements | On the operation day (Day 0)
  Aspartate aminotransferase (AST) in IU/L of participants was recorded from hospital's
Biochemical Measurements | On the operation day (Day 0)
  C-reactive protein (CRP) in mg/L of participants was recorded from hospital's patients form.
Biochemical Measurements | 7th day after the operation
  Albumin levels in g/dL of participants was recorded from hospital's patients form.
Biochemical Measurements | 7th day after the operation
  Prealbumin levels in mg/dL of participants was recorded from hospital's patients form.
Biochemical Measurements | 7th day after the operation
  Fasting Plasma glucose (FPG) mg/dL in of participants was recorded from hospital's patients form.
Biochemical Measurements | 7th day after the operation
  Alanine aminotransferase (ALT) in IU/L of participants was recorded from hospital's patients form.
Biochemical Measurements | 7th day after the operation
  Aspartate aminotransferase (AST) in IU/L of participants was recorded from hospital's patients form.
Biochemical Measurements | 7th day after the operation
  C-reactive protein (CRP) in mg/L of participants was recorded from hospital's patients form.

SECONDARY OUTCOMES:
Postoperative Complications of Participants | After the operation, up to 30 days.
  Infections (such as urinary tract, wound infections) and complications were recorded during the postoperative period.
Lenght of Hospital Stay of Participants | After the operation, up to 30 days.
  The length of patients' hospital stay were recorded during the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: BEDRİYE URAL, Dr, Principal Investigator — Saglik Bilimleri Universitesi; Elvan YILMAZ AKYUZ, Assoc. Prof., Principal Investigator — Saglik Bilimleri Universitesi; Cebrail AKYUZ, Assoc. Prof., Principal Investigator — Haydarpasa Numune Research and Training Hospital
Locations (1):
- Sağlık Bilimleri University, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fukatsu K. Role of nutrition in gastroenterological surgery. Ann Gastroenterol Surg. 2019 Feb 25;3(2):160-168. doi: 10.1002/ags3.12237. eCollection 2019 Mar. PMID 30923785
- [Background] Karimian J, Hadi A, Salehi-Sahlabadi A, Kafeshani M. The Effect of Arginine Intake on Colorectal Cancer: a Systematic Review of Literatures. Clin Nutr Res. 2019 Jul 25;8(3):209-218. doi: 10.7762/cnr.2019.8.3.209. eCollection 2019 Jul. PMID 31384599
- [Background] Bharadwaj S, Trivax B, Tandon P, Alkam B, Hanouneh I, Steiger E. Should perioperative immunonutrition for elective surgery be the current standard of care? Gastroenterol Rep (Oxf). 2016 May;4(2):87-95. doi: 10.1093/gastro/gow008. Epub 2016 Apr 14. PMID 27081153
- [Background] Moya P, Soriano-Irigaray L, Ramirez JM, Garcea A, Blasco O, Blanco FJ, Brugiotti C, Miranda E, Arroyo A. Perioperative Standard Oral Nutrition Supplements Versus Immunonutrition in Patients Undergoing Colorectal Resection in an Enhanced Recovery (ERAS) Protocol: A Multicenter Randomized Clinical Trial (SONVI Study). Medicine (Baltimore). 2016 May;95(21):e3704. doi: 10.1097/MD.0000000000003704. PMID 27227930
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Derived] Ural B, Yilmaz-Akyuz E, Akyuz C. Impact of Immunonutrition on Nutritional Status in Patients Undergoing Colorectal Cancer Surgery: A Randomized Controlled Clinical Trial. Nutr Cancer. 2024;76(6):469-475. doi: 10.1080/01635581.2024.2338607. Epub 2024 Apr 13. PMID 38613322